CLINICAL TRIAL: NCT02479594
Title: The Importance of Competence-feedback for Therapy Outcome: a Randomized Controlled Trial
Brief Title: Competence-feedback and Therapy Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University of Potsdam (Other)
Responsible Party: Principal Investigator, Florian Weck, Director of studies, University of Potsdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WE_01; WE 4652/7-1 (Other Grant/Funding Number: German Research foundation)
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Depression
Keywords: competence-feedback
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- competence-feedback (Experimental): Therapists assigned to this group will receive standardized feedback on their psychotherapeutic competency after every fourth treatment session with a patient for a period of 20 therapy sessions. The feedback will be given by two experienced raters who are licensed as psychological psychotherapists.
  Interventions: Behavioral: competence-feedback
- control (Placebo Comparator): Therapists assigned to this group will receive no competence-feedback.
  Interventions: Other: control

INTERVENTIONS:
Behavioral: competence-feedback — competence-feedback
  Arms: competence-feedback
Other: control — control group without competence-feedback
  Arms: control

SUMMARY:
In a randomized controlled study design, n = 58 treatments of patients with depression were to be conducted under a feedback-condition, in which the therapist would receive feedback five times within 20 treatment sessions. The competence-feedback includes detailed feedback about 14 different aspects of therapist behavior. The control group includes n = 58 further treatments within which therapists do not receive any competence-feedback (treatment as usual; TAU).

DETAILED DESCRIPTION:
Psychotherapeutic competencies are considered to be an important factor for therapy success. However, empirical studies which have investigated the competence-outcome relationship were only based on correlational analyses. Therefore, these studies are inappropriate for the investigation of causal relationships. In previous studies, feedback on therapists' competencies was found to be suitable for enhancing such competencies. Therefore, in the current research project, competence-feedback should be used to enhance therapeutic competencies systematically, in order to investigate the causal impact of these competencies on therapy outcome. Using a randomized controlled study design, n = 58 treatments of patients with depression were to be conducted under a feedback-condition, in which the therapist would receive feedback five times within 20 treatment sessions. The competence-feedback includes detailed feedback about 14 different aspects of therapist behavior. The control group includes n = 58 further treatments within which therapists do not receive any competence-feedback (treatment as usual; TAU). In order to ensure comparability of both treatment conditions (regarding an observation situation), the therapists in the TAU condition should also receive feedback, but only after the treatments are finished. We hypothesize that the feedback-group is superior to the TAU-group and that their treatments lead to significantly better therapy outcome. Moreover, we use mediator analysis to analyze whether the group-outcome relationship is mediated by therapeutic competencies or by the quality of the therapeutic alliance. The results are highly relevant for clinical process research, psychotherapy training and for the dissemination of treatment approaches in routine care.

ELIGIBILITY:
THERAPISTS

Inclusion Criteria:

* Having successfully completed the interim Audit
* Having started to treat ambulant patients

Exclusion Criteria:

---

PATIENTS

Inclusion Criteria:

* Clinical diagnosis of Major Depression (Meeting DSM-IV criteria)
* Informed consent

Exclusion Criteria:

* Suicidal tendency
* Clinical diagnosis of alcohol or drug addiction, acute schizophrenia, schizoaffective disorder or bipolar disorder
* Clinical diagnosis of personality disorder cluster A (odd disorders) and B (dramatic, emotional or erratic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-08; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory II (BDI II) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess depressive symptoms

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAMD-17) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  external assessment to assess depressive symptoms
Inventory of Interpersonal Problems (IIP-C) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report instrument to identify a person's salient interpersonal difficulties based on the interpersonal circumplex model
Health-related quality of life (SF-12) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess health-related quality of life
Client Satisfaction Questionaire (CSQ8) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess satisfaction with therapy
Cognitive Therapy Scale (CTS) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  external-assessment measure that assesses psychotherapeutic competency during a cognitive therapy session. CTS will be used by two trained raters licensed as psychological psychotherapists
Helping Alliance Questionaire (HAQ) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  self-report measure to assess therapeutic alliance from the therapists perspective (therapist version; HAQ-T), the patients perspective (HAQ-P) and the raters perspective (HAQ-R)
Assessment of Patient Interpersonal Behavior (AFPIB) | participants will be followed for the duration of psychotherapy, an expected average of 20 weeks
  assessment of patient in-session interpersonal behavior

CONTACTS AND LOCATIONS:
Overall Officials: Florian Weck, PhD, Study Director — University of Potsdam
Locations (1):
- Johannes Gutenberg University, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maass U, Witthoft M, Junga YM, Hahn D, Weck F. Relationships Among Patients' Interpersonal Behaviors in Sessions, Therapist Competence, and the Therapeutic Alliance in Cognitive Behavior Therapy: A Cross-Lagged Panel Analysis. J Clin Psychol. 2026 Jan;82(1):18-30. doi: 10.1002/jclp.70040. Epub 2025 Aug 30. PMID 40884452
- [Derived] Weck F, Junga YM, Kliegl R, Hahn D, Brucker K, Witthoft M. Effects of competence feedback on therapist competence and patient outcome: A randomized controlled trial. J Consult Clin Psychol. 2021 Nov;89(11):885-897. doi: 10.1037/ccp0000686. PMID 34881909